CLINICAL TRIAL: NCT03983473
Title: Identification of Fecal Microbiota Biomarkers of Spondyloarthritis in Patients Suffering From Crohn's Disease. Identification de Biomarqueurs de SPondylArthrite Chez Les Patients Atteints de Maladie de CROhn présents Dans le MICrobiote fécal.
Brief Title: Identification of Fecal Microbiota Biomarkers of Spondyloarthritis in Patients Suffering From Crohn's Disease.
Acronym: MICROSPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier Régional Metz-Thionville (Other); University Hospital, Strasbourg, France (Other); Saint Antoine University Hospital (Other)
Responsible Party: Principal Investigator, FERRY Marine, Doctor, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-A02298-31
Record Dates: First submitted 2019-05-22; First posted 2019-06-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease; Spondyloarthritis
MeSH Terms: conditions — Crohn Disease; Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Crohn's disease (Other): Patients suffering from established Crohn 's disease without spondyloarthritis
  Interventions: Other: Microbiota Sequencing
- Spondyloarthritis (Other): Patients with established spondyloarthritis without Crohn 's disease
  Interventions: Other: Microbiota Sequencing
- Crohn + spondyloarthritis (Other): Patients suffering from both spondyloarthritis and Crohn 's disease
  Interventions: Other: Microbiota Sequencing
- Healthy controls (Other): Patients without spondyloarthritis and Crohn 's disease
  Interventions: Other: Microbiota Sequencing

INTERVENTIONS:
Other: Microbiota Sequencing — virome, bacteriome, fungome NGS sequencing

SUMMARY:
The MICROSPA project aims to compare gut microbiota, serum cytokines, and PBMC of patients suffering from Crohn's disease (CD) associated or not to spondylarthritis (SpA). 3 groups of patients will be analyzed: patients suffering from CD alone, patients suffering from SpA alone, patients suffering from CD and SpA. One group of healthy controls will be analysed as a comparator. Fecal microbiota will be determined by bacteriome, virome and fungome NGS sequencing

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients will be recruited according to 3 groups:
* Patients with Crohn's disease and axial spondyloarthritis according to the criteria below.
* Patients with Crohn's disease (MC patients) with a diagnosis established according to clinical, biological criteria, radiological, endoscopic and / or histological studies for 3 months. With diagnosis of exclusion of a spondyloarthritis on criteria ASAS and / or New York modified.
* Patients with axial spondyloarthritis (SpA patients) with a diagnosis based on modified ASAS and / or New York criteria with exclusion diagnosis of Crohn's disease.
* Patient with the ability to give free and express informed consent.

Exclusion Criteria:

* History of colonic resection
* Taking antibiotics or colon preparation for colonoscopy within 8 weeks before stool collection (Temporary contraindication = removal possible before colic or first bowel preparation after the start of colonic preparation).
* Ostomy at the time of sampling
* BMI> 30
* extreme diet
* unbalanced diabetes
* Pregnant woman
* Patient under guardianship, under curatorship or under the protection of justice Contacts/Locations Central Contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-11-04 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Alpha and Beta diversity of Fecal bacteriome | + 6 months
  Alpha (number of species) and Beta diversity (distribution of species)
Alpha and Beta diversity of Fecal fungome | + 6 months
  Alpha (number of species) and Beta diversity (distribution of species)
Alpha and Beta diversity of Fecal virome | + 6 months
  Alpha (number of species) and Beta diversity (distribution of species)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Central Hospital, Nancy, Lorraine
  - Saint Antoine Hospital, Paris